CLINICAL TRIAL: NCT04825938
Title: Phase II Trial of Toripalimab, an Anti-PD-1 Monoclonal Antibody, in Combination With Combination Carboplatin and Nab-paclitaxel , as a Novel Neoadjuvant Pre-Surgical Therapy for Salivary Gland Malignant Neoplasms
Brief Title: Neoadjuvant Toripalimab in Combination With Carboplatin and Nab-paclitaxel in Untreated Salivary Gland Malignant Neoplasms
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Song Fan, MD, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Salivary Gland Malignant Neoplasms; Salivary Gland Tumors
MeSH Terms: interventions — toripalimab; Carboplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab + Carboplatin + Nab-paclitaxel (Experimental): * Toripalimab (IV), dose= 240mg , day=1 , cycle length: 21 days.
  * Carboplatin (IV), dose=300mg/m2, day= 1, cycle length: 21 days.
  * Nab-paclitaxel (IV), dose=260mg/m2, day= 1, cycle length: 21 days.
  Interventions: Drug: Toripalimab , Carboplatin, Nab-paclitaxel

INTERVENTIONS:
Drug: Toripalimab , Carboplatin, Nab-paclitaxel — Patients receive toripalimab IV on day 1, paclitaxel IV on day 1 and carboplatin IV on day 1 . Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

SUMMARY:
This proposed study will evaluate the efficacy and safety of preoperative administration Toripalimab combined with nab-paclitaxel and carboplatin in salivary gland malignant neoplasms who are about to undergo surgery.Monoclonal antibodies, such as Toripalimab , may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.This trial will be helpful for comprehensive exploratory characterization of tumor immune microenvironment and circulating immune cells in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of salivary gland cancers which is planned for treatment with curative intent including surgical resection: mucoepidermoid carcinoma, adenocarcinoma, adenoidcystic carcinoma, acinic cell carcinoma, or other histology .
* Greater than or equal to 18 and less than 80 years of age at time of study entry.
* ECOG performance status of 0 or 1.
* Measurable disease as per RECIST 1.1.
* Patients must have no prior exposure to immune-mediated therapy, including anti- cytotoxic T-lymphocyte protein 4 (CTLA-4), anti-programmed cell death 1, anti-programmed cell death 1 ligand 1 (PD-L1), or anti-programmed cell death ligand 2 antibodies, excluding therapeutic anticancer vaccines.
* Screening labs must meet the following criteria and must be obtained within 14 days prior to registration:

  1. Adequate hepatic and renal function as demonstrated by

     1. Serum creatinine < 1.5 X ULN or CrCl > 40mL/min (if using the Cockcroft-Gault formula below):

        * Males: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL)）
        * Females: Creatinine CL (mL/min) = (Weight (kg) x (140 - Age))/(72 x serum creatinine (mg/dL))x 0.85
     2. AST/ALT ≤ 3 x ULN
     3. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  2. Adequate bone marrow function as demonstrated by:

     1. Absolute Neutrophil Count >1,500/µL
     2. Platelets > 100 X 103/µL
     3. Hemoglobin > 9.0 g/dL
* Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 21 days of study enrollment.
* Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 23 weeks after the last dose of study drugs; "women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
* Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year; men who are receiving the study medications will be instructed to adhere to contraception for 31 weeks after the last dose of study drugs; men who are azoospermic do not require contraception.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Subjects must agree to allow use of any pre-treatment tissue remaining after definitive diagnosis is made (ie, archival and or fresh tissue) for research purposes. In addition, subjects must consent to allow use of their residual post-operative tissue for research purposes.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had another known invasive malignancy within the previous 5 years and/or has had surgery, chemotherapy, targeted small molecule therapy or radiation therapy within 5 years for a known malignancy prior to study day 0.
* If subject received major surgery for any other reason, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of day -5. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Has an active autoimmune disease requiring systemic steroid treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids.
* Active, known or suspected autoimmune disease. Note: Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger .
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* A history of allergic reaction attributed to compounds of similar chemical or biologic composition to the treatment or other agents used in the study.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibodies).
* Has known active Hepatitis B or C.
* Known history of active TB ( bacillus tuberculosis ).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events graded by CTCAE v5.0 | 90 days after the first dose of study treatment
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).
Percentage of participants demonstrating pathological response | At time of surgery
  Pathologic response in the primary tumor was assessed using a quantitative grading scheme:
  pathologic tumor response [nonviable tumor] PTR0 = no or <10% PTR1 = ≥10% PTR2 = ≥50%

SECONDARY OUTCOMES:
Disease-free survival （DFS） | 2 years
  DFS is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease relapse.
Overall survival（OS） | 5 years
  Overall survival will be defined as the time from day 1 of study treatment until death from any cause.
Radiographic Response | 5 weeks
  Radiographic response to treatment as defined by RECIST 1.1.
Pathologic Response | 6 weeks
  Pathologic response to neoadjuvant treatment in resected tumor and lymph nodes. The rate of major pathologic response, defined as <10% residual viable tumor cells in the resection specimen will be compared to historic data with neoadjuvant chemotherapy
Rate of surgery delay | 8 weeks after the patient receives their last dose
  Rate of patients with an Unplanned Delay to Surgery defined as any change to scheduled surgery date considered to be at least possibly related to neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China